CLINICAL TRIAL: NCT02200133
Title: Randomized Study of Individualized Care Plans for Hematopoietic Cell Transplant Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: Patient-Centered Outcomes Research Institute (Other); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-SCP
Record Dates: First submitted 2014-07-21; First posted 2014-07-25 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Adult Hematopoietic Cell Transplant (HCT) Survivors 1-2 Yrs Post Most Recent HCT
Keywords: Hematopoietic cell transplant (HCT) survivors; Survivorship Care Plan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized Survivorship Care Plan (SCP) (Experimental): * Participant information sheet and instructions on how to use the SCP
  * Patient version of individualized SCP that includes but is not limited to: (1) a treatment summary that consists of disease characteristics and treatment details (including HCT), and (2) recommendations for preventive care and screening for late complications based on patient treatment exposures (age, type of transplant, use of TBI, corticosteroid exposure as part of HCT, and history of GVHD)
  * Newest Vital Sign nutrition label to measure health literacy and its instructions
  * Participants may receive other materials their transplant center routinely provides to patients for follow-up care (e.g., discharge summary or clinic note)
  Interventions: Other: Individualized Survivorship Care Plan (SCP)
- Usual care (no SCP) (No Intervention): * Materials that their transplant center routinely provides to patients for follow-up care
  * Newest Vital Sign nutrition label to measure health literacy and its instructions
  * Participants randomized to the usual care arm who complete the 6 month study assessments will receive their individualized SCP upon completion of the patient's participation. Participants who withdraw from the study or who do not complete the 6 month assessment will not receive the individualized SCP.

INTERVENTIONS:
Other: Individualized Survivorship Care Plan (SCP) — The individualized SCP incorporates patient specific treatment exposures and provides a framework for long term followup based on those exposures and subsequent risks for late complications.
  Arms: Individualized Survivorship Care Plan (SCP)

SUMMARY:
This randomized study will compare a personalized Survivorship Care Plan (SCP) template with usual care (no SCP). The investigators hypothesize that the personalized SCP that incorporates patient specific treatment exposures and provides a framework for long term followup based on those exposures and subsequent risks for late complications will enhance patient survivorship confidence in knowledge, increase adherence to recommended healthcare, improve health behaviors and reduce HCT-related emotional distress.

DETAILED DESCRIPTION:
This randomized study will compare a personalized Survivorship Care Plan (SCP) template with usual care (no SCP). The investigators hypothesize that the personalized SCP that incorporates patient specific treatment exposures and provides a framework for long term followup based on those exposures and subsequent risks for late complications will enhance patient survivorship confidence in knowledge, increase adherence to recommended healthcare, improve health behaviors and reduce hematopoietic cell transplant (HCT) - related emotional distress.

The randomized study design will be able to evaluate the efficacy of individualized SCP in enhancing transplant survivor knowledge, health behaviors and health care utilization for recommended preventive care. Most transplant centers do not use a standardized SCP for their HCT recipients, and hence, the control arm would represent prevalent standard of care (e.g., discharge summary, provider-to-provider communication).

Transplant centers that will participate in this study will represent a spectrum of center types (e.g., geographic location, center volume, resources and infrastructure) and patient populations (e.g., healthcare disparities, urban/rural population, distance from transplant center). Usual care for each center will be documented at the time of determining center eligibility. The study principal investigators, in consultation with the protocol team, will make the determination about center eligibility after reviewing the centers "usual care" procedures. In order to avoid contamination of the study intervention, centers will be asked not to change their follow-up practices for the period they are enrolling patients on the study.

The primary objective of the investigators study is to evaluate the impact of an individualized SCP on survivor knowledge about past diagnostic and treatment details, confidence in knowledge about prevention and treatment of late-effects, access to resources and familial risk of cancer. For this objective, the investigators will compare the change in score on the Confidence in Survivorship Information instrument from baseline to 6 months after the study intervention.

Secondary objectives will investigate the influence of individualized SCP on standardized measures of HCT related distress, knowledge of recommended care, health behaviors, self-efficacy, and health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years at time of allogeneic HCT recipient at participating transplant centers)
* Survival 1-2 years after most recent HCT with no evidence of relapse, disease progression, or secondary cancer on last follow-up
* All diagnoses will be eligible
* All transplant types will be eligible (autologous or allogeneic related or unrelated)
* All graft sources will be eligible (bone marrow, peripheral blood or umbilical cord blood)
* All conditioning regimens will be eligible (in case of allogeneic HCT, patient could have received myeloablative or non-myeloablative/reduced-intensity conditioning)
* Patient may have received more than one HCT
* Patient must be proficient in English (written and spoken) to complete study assessments
* Patient must have a valid mailing address within the United States to receive study materials
* Signed informed consent form from patient

Exclusion Criteria:

- Patients who have received their transplant at a different transplant center will not be eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in Confidence in Survivorship Information instrument score | baseline to 6 months after the study intervention

SECONDARY OUTCOMES:
Change in HCT treatment distress instrument score | baseline to 6 months after the study intervention
Change in Health behaviors instrument score | baseline to 6 months after the study intervention
Changes in Healthcare utilization instrument score | baseline to 6 months after the study intervention
Change in Knowledge about transplant exposures instrument score | baseline to 6 months after the study intervention
Change in Quality of life instrument score | baseline to 6 months after the study intervention
Change in Self-efficacy instrument score | baseline to 6 months after the study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Murphy, EdD, RN, Study Chair — National Marrow Donor Program; Navneet Majhail, MD, MS, Study Chair — Cleveland Clinic Foundation; National Marrow Donor Program; K Scott Baker, MD, MS, Study Chair — Fred Hutchinson Cancer Center
Locations (17):
- United States (17):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Florida, Shands Hospital, Gainesville, Florida
  - Loyola Medical Center, Maywood, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington